CLINICAL TRIAL: NCT00163332
Title: Comparison of Inhaled Ciclesonide (160 mcg b.i.d. or 320 mcg b.i.d.) and Fluticasone Propionate (250 mcg b.i.d. or 500 mcg b.i.d.) in Pretreated Patients With Mild to Moderate Asthma
Brief Title: Effect of Inhaled Ciclesonide Versus Fluticasone Propionate in Patients With Mild to Moderate Asthma (18 to 65 y) (BY9010/M1-129)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BY9010/M1-129
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-09

CONDITIONS: Asthma
Keywords: Asthma; Ciclesonide; Fluticasone propionate
MeSH Terms: conditions — Asthma | interventions — ciclesonide

INTERVENTIONS:
Drug: Ciclesonide

SUMMARY:
The aim of the study is to investigate the effect of ciclesonide versus fluticasone propionate versus placebo on airway hyperresponsiveness and on the hypothalamic-pituitary-adrenal axis (HPA axis). Treatment medication will be administered as follows: ciclesonide or fluticasone propionate will be inhaled twice daily, using one of the two dose levels. The study duration consists of a baseline period (4 to 6 weeks), five treatment periods (9 days each), and a washout period between treatments (4 to 12 weeks). The study will provide further data on safety and tolerability of ciclesonide.

ELIGIBILITY:
Main Inclusion Criteria:

* Patients who have had a history of bronchial asthma for at least 6 months
* FEV1 >60% of predicted for at least 24 h
* Patients who are hyperresponsive to methacholine and to AMP
* Patients who are in good health with the exception of asthma

Main Exclusion Criteria:

* Concomitant severe diseases or diseases which are contraindications for the use of inhaled steroids
* Patients suffering from COPD and/or other relevant lung diseases except asthma
* Current smokers and ex-smokers both with ≥10 pack years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2003-03

PRIMARY OUTCOMES:
AUC(0-24h)/24 h of serum cortisol level
24 h urinary cortisol excretion adjusted for creatinine.

SECONDARY OUTCOMES:
8 am measurement of bone formation markers
PC20FEV1 to methacholine
PC20FEV1 to AMP
lung function (FEV1, FVC)
pharmacokinetics
safety and tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (5):
- Belgium (5):
  - Altana Pharma/Nycomed, Genk
  - Altana Pharma/Nycomed, Ghent
  - Altana Pharma/Nycomed, Lanaken
  - Altana Pharma/Nycomed, Liège
  - Altana Pharma/Nycomed, Liége

REFERENCES:
- See also: BY9010-MI-129-RDS-2007-04-25.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4517&filename=BY9010-MI-129-RDS-2007-04-25.pdf